CLINICAL TRIAL: NCT07339800
Title: Chest CT Scan in Pulmonary Mucormycosis: Prognostic Value
Acronym: RadioMucor
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9767
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Mucormycosis
Keywords: Pulmonary Mucormycosis; Fungal infections
MeSH Terms: conditions — Mycoses

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Invasive pulmonary fungal infections caused by Mucorales are rare but severe and rapidly progressive, affecting immunocompromised patients. The role of chest imaging in their diagnosis is well established in the 2020 EORTC/MSGERC criteria, and its use is almost systematic. However, the progression of lung parenchymal involvement and any potential prognostic radiological patterns in the follow-up of these infections are less well understood. This research aims to identify imaging characteristics predictive of favorable or unfavorable outcomes in infected patients, in order to better tailor follow-up and therapeutic options.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Treated at Strasbourg University Hospital between January 1, 2009, and June 3, 2025
* With a diagnosis of probable or proven invasive pulmonary infection with Mucorales according to the 2020 EORTC/MSGERC criteria
* Having undergone at least one CT scan including the thoracic region

Exclusion Criteria:

* No CT scan including the thoracic region
* No diagnosis of probable or proven invasive pulmonary infection with Mucorales (EORTC/MSGERC 2020 criteria)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a diagnosis of probable or proven invasive pulmonary infection with Mucorales according to the 2020 EORTC/MSGERC criteria
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-09-18 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09-19 (Estimated)

PRIMARY OUTCOMES:
Death rate in patients with probable or proven invasive Mucorales infection | Day 15 after infection
  Death rate at day 15 in patients with probable or proven invasive Mucorales infection

CONTACTS AND LOCATIONS:
Locations (1):
- Service des Maladies Infectieuses et Tropicales - CHU de Strasbourg - France, Strasbourg, France